CLINICAL TRIAL: NCT00230633
Title: Studies of White Blood Cells Derived From HHT Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS3
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Telangiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with HHT: People with molecularly confirmed HHT. No intervention, blood sample only
- Controls: People without HHT No intervention, blood sample only

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT, also known as Osler-Weber-Rendu Syndrome) is an inherited vascular disease that leads to the development of dilated and fragile blood vessels. The study goal is to culture white blood cells that express the proteins mutated in HHT and examine in the laboratory to explain aspects of the HHT disease phenotype.

DETAILED DESCRIPTION:
HHT is a vascular condition but many of the genes that are mutated to cause HHT (endoglin, ALK-1 and SMAD4) are also expressed in white blood cells. In this study, investigators will take blood samples from people with HHT, culture the white blood cells and study their properties in media prompting different types of differentiation, or infection of cell lines with Epstein Barr virus to provide cell lines which can be repeatedly studied. RNA and proteins will be extracted from these cells for study of white cell responses and association with expression levels of endoglin, ALK-1 and SMAD4. The investigators hypothesize that these cells which express "half-normal" endoglin, ALK-1 or SMAD4 will show differences when compared to normal white blood cells. It is also anticipated that that these findings may help to explain aspects of the HHT disease phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HHT,
* HHT patients family members

Exclusion Criteria:

* Unable to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hereditary hemorrhagic telangiectasia (HHT) and controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-04 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Proteins and cellular markers related to coagulation | on average completing each biomarker study in 1-5 years
  Not specified at outset. Blood samples will be collected over the recruitment period, usually on a single day. Analyses of biomarkers relate to the SAME DAY, within 24hs, though will be evaluated over subsequent months, on average completing in 1-5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom

REFERENCES:
- [Background] Clarke JM, Alikian M, Xiao S, Kasperaviciute D, Thomas E, Turbin I, Olupona K, Cifra E, Curetean E, Ferguson T, Redhead J; Genomics England Research Consortium; Shovlin CL. Low grade mosaicism in hereditary haemorrhagic telangiectasia identified by bidirectional whole genome sequencing reads through the 100,000 Genomes Project clinical diagnostic pipeline. J Med Genet. 2020 Dec;57(12):859-862. doi: 10.1136/jmedgenet-2019-106794. Epub 2020 Apr 17. No abstract available. PMID 32303606
- [Background] Balachandar S, Graves TJ, Shimonty A, Kerr K, Kilner J, Xiao S, Slade R, Sroya M, Alikian M, Curetean E, Thomas E, McConnell VPM, McKee S, Boardman-Pretty F, Devereau A, Fowler TA, Caulfield MJ, Alton EW, Ferguson T, Redhead J, McKnight AJ, Thomas GA; Genomics England Research Consortium; Aldred MA, Shovlin CL. Identification and validation of a novel pathogenic variant in GDF2 (BMP9) responsible for hereditary hemorrhagic telangiectasia and pulmonary arteriovenous malformations. Am J Med Genet A. 2022 Mar;188(3):959-964. doi: 10.1002/ajmg.a.62584. Epub 2021 Dec 13. PMID 34904380
- [Result] Shovlin CL, Sulaiman NL, Govani FS, Jackson JE, Begbie ME. Elevated factor VIII in hereditary haemorrhagic telangiectasia (HHT): association with venous thromboembolism. Thromb Haemost. 2007 Nov;98(5):1031-9. PMID 18000608
- [Result] Shovlin CL, Chamali B, Santhirapala V, Livesey JA, Angus G, Manning R, Laffan MA, Meek J, Tighe HC, Jackson JE. Ischaemic strokes in patients with pulmonary arteriovenous malformations and hereditary hemorrhagic telangiectasia: associations with iron deficiency and platelets. PLoS One. 2014 Feb 19;9(2):e88812. doi: 10.1371/journal.pone.0088812. eCollection 2014. PMID 24586400